CLINICAL TRIAL: NCT01107366
Title: Extensive Type A Dissections and Thoracic/ Thoraco-Abdominal
Brief Title: ATLANTIS:Extensive Type A Dissections and Thoracic/ Thoraco-Abdominal Aneurysms Repair With LupiAe Hybrid TechNique
Acronym: ATLANTIS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study never started since our Medical Ethic Commeettee did not approved it
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: prof roberto di bartolomeo, cardiochirurgia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATLANTIS BOLOGNA
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Aortic Aneurysm
Keywords: lupiae techinque; aortic aneurism; aortic dissection
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: lupiae technique — it's a new hybrid technique for the treatment of aortic aneurism and dissection.
Procedure: lupiae technique — LUPIAE technique
  Hybrid repair of thoracic or thoraco-abdominal aneurysms of different etiology and type A dissections with a two-stage procedure:
  1. surgical arch reconstruction with a Dacron multibranched surgical prothesis
  2. endovascular implantation of a thoracic stent graft

SUMMARY:
To prospectively evaluate the safety and efficacy of the LUPIAE hybrid technique for the treatment of

* thoracic or thoraco-abdominal aortic aneurysms
* thoracic aortic type A dissections 2. to compare the safety and efficacy of the LUPIAE hybrid technique with historical groups (literature review, other hybrid techniques, LUPIAE retrospective patients)

DETAILED DESCRIPTION:
LUPIAE technique:

Hybrid repair of thoracic or thoraco-abdominal aneurysms of different etiology and type A dissections with a two-stage procedure:

1. surgical arch reconstruction with a Dacron multibranched surgical prothesis
2. endovascular implantation of a thoracic stent graft

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing to sign the informed consent, or In case of acute patients that should arrive at the hospital in unconsciousness status, patient's first degree relatives willingness to sign the informed consent and patient's willingness to re-consent for the study participation once he/she is again conscious.

   and
2. Patients with extensive thoracic or thoraco-abdominal aortic aneurysms (>55 mm diameter), involving the ascending, arch and descending aortic segments, but not involving the renal arteries (at least 15 mm of healthy tissue above the most proximal renal artery).

   Or
3. Patients with extensive type A aortic dissection (DeBakey type I) with at least one of the following minimum criteria:

   * An initial false lumen diameter measured in the upper descending thoracic aorta >22 mm;
   * Total aortic diameter measured in the descending thoracic aorta >45 mm;
   * True lumen's compression (True lumen <10% of total aortic lumen);
   * Non-controlled hypertension;
   * Persistent pain;
   * Rupture or imminent rupture;

Exclusion Criteria:

1. Patient has a standard contraindication to the implant of thoracic stent graft;
2. Patient unable to commit to follow-up schedule;
3. Patient has medical conditions that preclude protocol required testing or limit study participation;
4. Patient is enrolled or intend to participate in another clinical trial during the course of this study;
5. Less than 18 years of age;
6. Pregnancy;
7. A life expectancy of less than one year, except for Patients with extensive type A aortic dissection (DeBakey type I)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico S Orsola Malpighi, Bologna, Italy, Italy